CLINICAL TRIAL: NCT00316979
Title: Therapeutic Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) in the Treatment of Migraine Using Somatosensory Evoked High-Frequency Oscillations as a Parameter: A 3-year Study.
Brief Title: Efficacy of rTMS in the Treatment of Patients With Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rTMS_Migraine_VGHTPE
Record Dates: First submitted 2006-04-20; First posted 2006-04-21 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Migraine
Keywords: migraine; transcranial magnetic stimulation; repetitive transcranial magnetic stimulation; rTMS
MeSH Terms: conditions — Migraine Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

SUMMARY:
Migraine is a condition thought to be related to cortical hyperexcitability. Repetitive transcranial magnetic stimulation (rTMS) can modulate the cortical excitability by means of long-term potentiation or long-term depression. This study will will test the safety and efficacy of rTMS in the treatment of patients with Migraine.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-65 years
* Diagnosed as migraine (with or without aura)
* More than 4 attacks per month for at least 3 months prior to study
* No preventive medication used
* Must be able to sign permit

Exclusion Criteria:

* History of seizure or family history of seizures
* Women in pregnancy or breast-feeding
* Patient with medication overuse
* Patient with other medical, psychologic, or surgical illness
* Patient under preventive medications
* Prior rTMS examination one month within

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2006-04

PRIMARY OUTCOMES:
Reduction in days of migraine attack per month

SECONDARY OUTCOMES:
The reduction in dosage of acute abortive medication
The reduction of headache index

CONTACTS AND LOCATIONS:
Overall Officials: Shuu-Jiun Wang, MD, Principal Investigator — Headache Center, Taipei Veterans General Hospital
Locations (1):
- Headache Center, Teipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Brighina F, Piazza A, Vitello G, Aloisio A, Palermo A, Daniele O, Fierro B. rTMS of the prefrontal cortex in the treatment of chronic migraine: a pilot study. J Neurol Sci. 2004 Dec 15;227(1):67-71. doi: 10.1016/j.jns.2004.08.008. PMID 15546593
- [Background] Lorenz J, Minoshima S, Casey KL. Keeping pain out of mind: the role of the dorsolateral prefrontal cortex in pain modulation. Brain. 2003 May;126(Pt 5):1079-91. doi: 10.1093/brain/awg102. PMID 12690048